CLINICAL TRIAL: NCT06684522
Title: Upadacitinib As a Novel Treatment for Refractory Eyelid Dermatitis
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Walter Liszewski, Principal Investigator, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00221561
Record Dates: First submitted 2024-11-10; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-10

CONDITIONS: Eyelid Dermatitis
MeSH Terms: interventions — upadacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Upadacitinib Treatment (Experimental): Participants on upadacitinib 15mg daily
  Interventions: Drug: Upadacitinib 15 MG

INTERVENTIONS:
Drug: Upadacitinib 15 MG — Upadacitinib 15mg daily
  Other Names: RINVOQ

SUMMARY:
This study aims to assess the efficacy of upadacitinib in eyelid dermatitis that has not resolved with topical therapies and patch testing.

ELIGIBILITY:
Inclusion Criteria:

* Individuals age 18-70 years old with eyelid dermatitis for at least two months
* Failure of at least one topical prescription cream for the eyelid dermatitis (steroid, pimecrolimus, tacrolimus, crisaborole, or ruxolitinib)
* Women of reproductive potential must agree to using effective contraception during treatment and for 4 weeks following the final dose of Upadacitinib.
* Willing and able participants that provide informed consent
* Willing and able participants that comply with study activities

Exclusion Criteria:

* Self-reported history of allergic response to upadacitinib
* Subject with self-reported history of heart disease, stroke, or neurological conditions
* Currently taking topical medications for eyelid dermatitis within one week of starting study drug
* Women who are pregnant, nursing, or who may become pregnant during the study
* Non-English-speaking subjects
* Patients with an active serious infection
* Patients with active TB or latent TB, patients should be tested for TB prior to upadacitinib treatment.
* Patients with active HBV/HCV or abnormal lab ranges, Lab Data: Hb<8g/dL, ALC<500 cells/mm3 and ANC <1000 cells/mm3
* Patients with a history of malignancy within the last 5 years other than successfully treated NMSC.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Reduction in Investigator Global Assessment (IGA) | 12 weeks
  Reduction in baseline IGA score at week 12 compared to week 0

CONTACTS AND LOCATIONS:
Overall Officials: Walter Liszewski, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Department of Dermatology, Chicago, Illinois, United States